CLINICAL TRIAL: NCT05449925
Title: Title: Effect Of Injectable Platelet Rich Fibrin With Microneedling On Thin Gingival Phenotype In Fixed Non Extraction Orthodontic Cases - A Randomized Controlled Clinical Trial
Brief Title: Effect Of Injectable PRF And Microneedling In Patient Undergoing Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mrinalini Verma Perio
Record Dates: First submitted 2022-05-30; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Thin-gingiva
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST GROUP (Experimental): i-PRF and Microneedling Procedure in thin gingiva followed by orthodontic treatment
  Interventions: Procedure: Injectable PRF and Microneedling
- CONTROL GROUP (No Intervention): no periodontal intervention

INTERVENTIONS:
Procedure: Injectable PRF and Microneedling — i-PRF and Microneedling Procedure in thin gingiva followed by orthodontic treatment
  Arms: TEST GROUP

SUMMARY:
To evaluate the effect injectable platelet rich fibrin (i-PRF) along with microneedling on gingival thickness in patients with thin gingival phenotype undergoing non extraction fixed orthodontic treatment

DETAILED DESCRIPTION:
A non surgical, non invasive method of increasing gingival thickness has been reported using injectable platelet rich fibrin (i-PRF) alone and with microneedling (MN) in individuals with thin periodontal phenotype .

I-PRF is prepared as per low speed centrifugation concept that can provide a significant advantage for the regeneration process as it is rich in platelets, leukocytes, growth factors (As iprf is rich in WBC'c enabling slow and sustained release of growth factors as it clots and forms a gel approximately after 10-15 min and preserve its contents in the tissue for sustained release and inducing the expression of transforming growth factor-β11 and collagen-1 mRNA11, cellular fibroblasts11 and osteoblasts migration10 and collagen-1 synthesis10 .

Microneedling (MN) is also called as "percutaneous collagen induction therapy"9. Microinjuries created by MN result in minimal superficial bleedings and create a wound healing cascade which includes neocollagenesis and neoangiogenesis from which various growth factors, such as platelet derived growth factors, transforming growth factors, connective tissue growth factor and fibroblast growth factors are released9.

Primary therapeutic goal of this study is to do preorthodontic gingival augmentation using a latest technique injectable platelet rich fibrin (iprf) along with microneedling (MN) to increase the buccolingual thickness of marginal tissues over teeth that creates more robust marginal tissues that are less susceptible to trauma or plaque related inflammation and subsequent recession.

AIM : The primary aim of the study is to evaluate the effect injectable platelet rich fibrin (i-PRF) along with microneedling on gingival thickness in patients with thin gingival phenotype undergoing non extraction fixed orthodontic treatment.

OBJECTIVES

PRIMARY OBJECTIVE :

1. To measure and compare gingival tissue thickness in mandibular anteriors in patients requiring labial orthodontic movement (in non extraction cases) with thin gingival phenotype by using injectable platelet rich fibrin and microneedling (TEST GROUP) without using injectable platelet rich fibrin and microneedling(CONTROL GROUP ).

SECONDARY OBJECTIVE :

1. To evaluate keratinized tissue width ( KTW ) in mandibular anteriors in patients requiring labial orthodontic movement without extraction by using injectable platelet rich fibrin (TEST GROUP) and without using injectable platelet rich fibrin(CONTROL GROUP ).
2. To measure and compare effect of microneedling and i-PRF on periodontal parameter PI,GI,BOP,PD,CAL in mandibular anteriors in patients requiring labial orthodontic movement in non extraction cases.

INTERVENTION

IN TEST GROUP :

Local anaesthesia in the form of xylocaine HCL (2%) will be administered. i-PRF Preparation : A venous blood sample will be taken once for each patient using a 20 ml injector will be separated into two PRF tubes of 10 ml each containing no anticoagulant and centrifuged at room temperature with choukron's protocol. The i-PRFs obtained will be placed in 2.5cc dental injectors. The 27-gauge dental injector needles will be used for injection of i-PRF.

Microneedling Procedure :

Thirty-gauge (0.255 mm) lancet needles will be vertically inserted into the tissue until the hard tissue will reach. MN will be carried out on keratinized gingiva from the mesial line of the central tooth to the distal part of the canine tooth to be treated with the help of a lancet.

After one week post scaling, sites will be treated with i-PRF and microneedling. A total of 4 sessions will be done with an interval of 10 days each.

IN CONTROL GROUP :

Patients undergoing orthodontic treatment for labial retraction of mandibular anteriors with thin gingival phenotype will be kept under observation for 6 months for gingival phenotype with follow up.

STUDY DESIGN AND SETTING The present prospective, analytical, randomized clinical trial, single blinded study was conducted in the Department of PERIODONTOLOGY, Post Graduate Institute Of Dental Sciences, Rohtak.

STUDY PERIOD MARCH 2021 to 2022 JULY FOLLOW UP 6 months STUDY SUBJECTS TEST GROUP = 18 CONTROL GROUP = 18

ELIGIBILITY:
Inclusion Criteria:

* • GT of the mandibular anterior teeth <1mm (jepson et al. 2018) requiring labial orthodontic tooth movement without extraction.

  * Patients with > 18 years who will be systemically healthy
  * full-mouth plaque index (PI) and full-mouth bleeding on probing (BOP) score of ≤ 15%
  * gingival index (GI) of <1 (loe and silness) and dehiscence in mandibular anterior teeth detected in CBCT;

Exclusion Criteria:

* Patients with thick gingival biotype (>1mm gingival thickness as per Jepson et al.,2018) ;
* Patient undergoing dental extraction for labial orthodontic tooth movement.
* previous periodontal surgery;
* systemic disease;
* smokers
* use of blood thinners;
* use of any drugs that might lead to gingival enlargement;
* mucogingival stress, bruxism.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-08-25 (Estimated)

PRIMARY OUTCOMES:
Change in Gingival tissue thickness (GTT) | 6 months
  Change in Gingival tissue thickness from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: MRINALINI VERMA, BDS, Principal Investigator — PGIDS, ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No